CLINICAL TRIAL: NCT02183792
Title: Aquaresis Utility for Hyponatremic Acute Heart Failure Study
Acronym: AQUA-AHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Tien Ng, Associate Professor of Clinical Pharmacy and Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-13-00705
Record Dates: First submitted 2014-06-25; First posted 2014-07-08 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental): Tolvaptan 30-60mg once daily (with rescue loop diuretic or metolazone)
  Interventions: Drug: Tolvaptan
- Furosemide (Active Comparator): Furosemide continuous infusion 5mg/h with option to titrate (with rescue metolazone)
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Tolvaptan
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Furosemide
  Other Names: Lasix
  Arms: Furosemide

SUMMARY:
Hyponatremia is a common finding in acute heart failure (HF) patients and is associated with worse prognosis. In addition to its prognostic value, hyponatremia may have importance during the acute management of HF. We've recently shown that acute or chronic hyponatremia, especially <130 mEq/L, was associated with higher loop diuretic dose requirements and more frequent need for escalation of the diuretic regimen to achieve the same level of diuresis as normonatremic HF patients. Aquaresis with tolvaptan represents a potentially advantageous approach to the management of volume overload in HF, especially in patients presenting with concomitant hyponatremia. The purpose of the current study is to prospectively evaluate the comparative efficacy and safety of a tolvaptan-based diuretic regimen compared to conventional diuresis with a furosemide-based regimen on short-term clinical and treatment outcomes in hyponatremic acute HF patients.

This will be a prospective, open-label, parallel-group, randomized study comparing a tolvaptan-based aquaretic regimen to a conventional continuous infusion loop diuretic-based regimen of furosemide. Up to 55 (target sample size of 50) adult subjects admitted with acute HF and signs of volume overload, and serum sodium less than 135 mEq/L will be randomized to tolvaptan or furosemide treatment arms. The initial 24 hours of study treatment will compare tolvaptan monotherapy to furosemide monotherapy. After the initial 24 hours, treatment regimens may be altered to achieve desired clinical goals. Patients will be followed for up to 96 hours and at discharge for study purposes.

ELIGIBILITY:
Inclusion Criteria:

* Acute HF with signs or symptoms of volume overload [i.e. elevated jugular venous pulsation (JVP), rales, edema]
* Serum sodium < 135 mEq/L at time of or within first 48 hours of hospitalization
* Randomized within 48 hours of presentation to hospital
* ≥ 18 years of age
* Informed consent

Exclusion Criteria:

* Severe symptomatic hyponatremia requiring acute treatment
* Severe renal impairment upon admission (creatinine clearance < 20 mL/min)
* Renal replacement therapy dependent, or requiring upon admission
* Acute coronary syndrome on admission
* Requires or has a mechanical circulatory support device
* Evidence of cardiogenic shock requiring intravenous vasopressors
* Pregnancy
* Patient requiring concomitant use of strong CYP3A4 inhibitors (clarithromycin, ketoconazole, itraconazole, ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, and telithromycin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tien Ng, PharmD, Principal Investigator — University of Southern California; Uri Elkayam, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Keck Medical Center of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolvaptan: Tolvaptan 30-60mg once daily (with rescue loop diuretic or metolazone)
  Tolvaptan
- Furosemide: Furosemide continuous infusion 5mg/h with option to titrate (with rescue metolazone)
  Furosemide
Period: Overall Study
Arm/Group | Tolvaptan | Furosemide
Started | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan | Furosemide | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.7) | 59 (8.9) | 56 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33
Home Loop Diuretic Dose (Furosemide equivalents) [Mean (Standard Deviation); unit: mg] | 93 (63.5) | 108 (77.5) | 100 (68.5)

OUTCOME MEASURES:

1. Primary Outcome: Median Urine Output at 24 Hours Post Randomization
Time Frame: 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tolvaptan | Furosemide
Number analyzed (Participants) | 18 | 15
mL | 2910 [1100 to 4225] | 3150 [2375 to 5680]

2. Secondary Outcome: Median Change in Serum Creatinine at 24 Hours Post Randomization
Description: Comparison between baseline and 24 hours post randomization concentrations.
Time Frame: 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tolvaptan | Furosemide
Number analyzed (Participants) | 18 | 15
mg/dL
  Median Scr at Baseline | 1.15 [0.88 to 1.51] | 0.87 [0.76 to 1.22]
  Median Scr at 24h | 1.06 [0.76 to 1.37] | 0.96 [-0.19 to 1.53]
  Median 24h Change | -0.08 [-0.14 to -0.04] | -0.01 [-0.19 to 0.15]

3. Other Pre Specified Outcome: Total Urine Output
Time Frame: Up to 96 hours post randomization and participants will be followed for the duration of hospital stay, an expected average of 5 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Glomerular Filtration Rate (Estimated)
Time Frame: as for outcome 3
Reporting Status: Not Posted

5. Other Pre Specified Outcome: In-hospital Mortality
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mean Hourly Urine Output at 24 Hours
Time Frame: as for outcome 3
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Serum Sodium Change
Description: Difference assessed at baseline, 8, 24, 48, 72 and 96 hours.
Time Frame: as for outcome 3
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Weight Change
Description: Difference assessed at baseline, 8, 24, 48, 72 and 96 hours.
Time Frame: as for outcome 3
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Cumulative Furosemide Dose
Time Frame: as for outcome 3
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Cumulative Metolazone Use
Time Frame: as for outcome 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Self-rated Dyspnea
Time Frame: At baseline, 24 and 96 hours post randomization
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Acute Worsening of Kidney Function (Defined as an Increase in Serum Creatinine 0.3 mg/dL or 25% Above Baseline)
Time Frame: as for outcome 3
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Incidence of Electrolyte Abnormalities
Description: Hypo- and hyperkalemia defined as outside the range of 3.5 to 5.0 mEq/L Hypo- and hypermagnesemia defined as outside the range of 1.5-2.4 mEq/L
Time Frame: as for outcome 3
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Symptomatic Hypotension
Time Frame: as for outcome 3
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Plasma Renin Activity
Time Frame: At baseline, 24 and 96 hours post randomization
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Copeptin
Time Frame: At baseline, 24 and 96 hours post randomization
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in N-terminal Pro-B-type Natriuretic Peptide
Time Frame: At baseline, 24 and 96 hours post randomization
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Cystatin C
Time Frame: At baseline, 24 and 96 hours post randomization
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Urinary Neutrophil Gelatinase-associated Lipocalin (NGAL)
Time Frame: At baseline, 24, 48, 72 and 96 hours post randomization
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Hospital Length of Stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During hospitalization (up to 96 hours post randomization)
Arm/Group | Tolvaptan | Furosemide
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02183792/Prot_SAP_000.pdf